CLINICAL TRIAL: NCT01968447
Title: Effect of Deep Neuromuscular Block and Variations in Arterial PCO2 on the Surgical Rating Scale (SRS), Extubation Conditions and Postoperative Conditions Following Reversal With Sugammadex
Brief Title: Effect of Neuromuscular Block and Arterial PCO2 on Surgical Rating Scale (SRS), Following Reversal With Sugammadex
Acronym: BLISSS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Albert Dahan, Prof. Dr., Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL45461.058.13
Record Dates: First submitted 2013-10-07; First posted 2013-10-24 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-02

CONDITIONS: Prostate Cancer; Renal Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hypocapnia (Experimental): arterial pCO2 of 3.5 kPa
  Interventions: Other: hypocapnia
- normocapnia (Active Comparator): arterial PCO2 of 6.5-7.0 kPa
  Interventions: Other: normocapnia

INTERVENTIONS:
Other: hypocapnia — Hyperventilation to the level of hypocapnia
  Other Names: Low CO2
  Arms: hypocapnia
Other: normocapnia — Normal ventilation to the level of nromocapnia
  Other Names: normal CO2
  Arms: normocapnia

SUMMARY:
The purpose of this study is to study the effect of variations in the arterial CO2 concentration during deep neuromuscular block on the surgical conditions as assessed by the surgical rating scale

DETAILED DESCRIPTION:
Surgical conditions in laparoscopic surgery are largely determined by the depth of neuromuscular relaxation during surgery. This is especially true in procedures which are confined to a narrow working field such as retroperitoneal laparoscopic surgery (eg. renal and prostatic surgery). In the previous study (BLISS study) deep neuromuscular block (NMB) has shown to provide superior surgical conditions compared to moderate NMB. Moreover, rapid reversal of a deep NMB at the end of surgery was possible with Sugammadex (4mg/kg). The deep NMB did not lead to any delay in extubation time and did not cause any prolongation of stay in the recovery room when the block was reversed with Sugammadex

Rapid, safe and complete reversal of profound NMB blockade was not possible until the discovery of Sugammadex. Sugammadex is a modified γ-cyclodextrin. It was developed to selectively bind free plasma rocuronium, a non-depolarizing steroidal neuromuscular blocking agent. The BLISS study was the first study in which the effect of deep NMB on surgical conditions was assessed. Surgical conditions in this study were scored by one surgeon on a newly applied surgical rating scale which ranges from one to five.

Although the BLISS study showed that a deep NMB provided better surgical conditions than a moderately deep NMB overall, there was a high variability in surgical rating scores. More over, even at the deep NMB, SRS scores of 3 (moderate, but acceptable conditions) were noted. This indicates that surgical conditions are influenced by other factors as well. Involuntary movement of the diaphragm is possibly such a major disturbant of the surgical field. Previous studies have shown a relative resistance to neuromuscular blocking agents of the diaphragm compared to the musclus adductor pollicis on which neuromuscular block is generally monitored. Hence contractions of the diaphragm may occure despite a deep NMB. This may be due to (high) arterial carbon dioxide (CO2) concentrations, which stimulate the respiratory neuronal pool in the brainstem and consequently activate the phrenic nerve. In normal circumstances, the respiratory centers try to maintain an arterial CO2 pressure of 40 mmHg. With intentional hyperventilation, the arterial CO2 pressure may be lowered to 10-20 mmHg. A low arterial CO2 pressure diminishes the respiratory drive and consequently phrenic nerve activity. This is supported by previous observations which showed increased abdominal muscle relaxation produced by hyperventilation. We therefore designed this study to evaluate the effect of arterial CO2 variation with concurrent deep NMB on the surgical conditions. Arterial CO2 tensions may be altered by adjusting the ventilator settings. Eg. by increasing minute ventilation volume, arterial CO2 concentration will lower. Regular arterial blood samples will be drawn to monitor arterial CO2 concentration.

We hypothesize that a Deep NMB combined with hypocapnia will result in a significant improvement of surgical conditions as rated on the surgical rating scale by one surgeon compared to deep NMB and normocapnia

Additional secondary end-points of the study include the effect of arterial CO2 variation on:

* economic parameters (time to spontaneous breathing, time to extubation, duration of surgery, and time in the post-anesthesia care unit)
* perioperative hemodynamics, abdominal pressure
* postoperative conditions (respiratory conditions, hemodynamics, arterial oxygen saturation, pain, sedation, nausea and vomiting)
* To assess the ability of anesthesiologists and surgeons to rate the surgical field using video snippets of the surgical field.

ELIGIBILITY:
Inclusion Criteria:

* (i) Patients diagnosed with renal or prostatic disease who are will undergo an elective laparoscopic renal surgical procedure or laparoscopic prostatectomy;
* (ii) ASA class I-III
* (iii) > 18 years of age;
* (iv) Ability to give oral and written informed consent.

Exclusion Criteria:

* (i) Known or suspected neuromuscular disorders impairing neuromuscular function;
* (ii) Allergies to muscle relaxants, anesthetics or narcotics;
* (iii) A (family) history of malignant hyperthermia;
* (iv) Women who are or may be pregnant or are currently breast feeding;
* (v) Renal insufficiency, as defined by serum creatinine x 2 of normal, or urine output < 0.5 ml/kg/h for at least 6 h. When available, other indices will be taken into account as well such as glomerular filtration rate < 60 ml/h and proteinuria (a ratio of 30 mg albumin to 1 g of creatinine).
* (vi) Previous retroperitoneal surgery at the site of the current surgery.
* (vii) Body mass index > 35 kg/m2
* (viii) Chronic obstructive pulmonary disease GOLD 2-4 or a FEV1 less than 70% predicted or VC less than 70% predicted
* (ix) chronic pulmonary disease with altered lung physiology (eg. sarcoidosis, cycstic fibrosis, obstructing pulmonary tumors, previous lung surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Dahan, MD, Principal Investigator — LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boon M, Martini C, Hellinga M, Bevers R, Aarts L, Dahan A. Influence of variations in arterial PCO2 on surgical conditions during laparoscopic retroperitoneal surgery. Br J Anaesth. 2016 Jul;117(1):59-65. doi: 10.1093/bja/aew114. Epub 2016 May 6. PMID 27154574

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypocapnia: arterial pCO2 of 3.5 kPa or 26.3 mmHg
  hypocapnia
- Normocapnia: arterial PCO2 of 6.5-7.0 kPa or 48.8-52.5 mmHg
  normocapnia
Period: Overall Study
Arm/Group | Hypocapnia | Normocapnia
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypocapnia | Normocapnia | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 10 | 8 | 18
Age, Continuous [Median (Full Range); unit: years] | 65 [22 to 80] | 62 [25 to 72] | 64 [22 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 17 | 14 | 31
Region of Enrollment [Number; unit: participants]
  Netherlands | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Surgical Rating Scale
Description: During a procedure, the surgical condition will be scored by one surgeon using a 5-point surgical rating scale. The rating scale is a 5-point ordinal scale ranging from 1 = poor condition to 5 = optimal surgical conditions. The surgeon will score the condition at 15 minute intervals.The values given on the surgical rating scale are averaged and the average value is used in the data analysis.
Time Frame: Peroperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypocapnia | Normocapnia
Number analyzed (Participants) | 20 | 20
units on a scale | 4.86 (0.4) | 4.75 (0.4)
Statistical Analysis 1: Comparison: Hypocapnia vs Normocapnia; Test type: Superiority or Other; p = 0.59, Mixed Models Analysis

2. Secondary Outcome: Hemodynamics
Description: Hemodynamic conditions are studied during low arterial CO2 concentration and normal arterial CO2 concentration. The average of the measured mean arterial pressures at 15 minute intervals during anesthesia are presented
Time Frame: peroperative
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Hypocapnia | Normocapnia
Number analyzed (Participants) | 20 | 20
millimeters of mercury | 85 (10) | 81 (9)

3. Secondary Outcome: Respiratory Function
Description: The effect of low versus normal pCO2 concentrations on the postoperative respiratory function will be studied. Postoperative saturations are obtained at 15 minutes intervals. The data are averaged over time.
Time Frame: from the end of surgery untill 2 hours postoperative
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Hypocapnia | Normocapnia
Number analyzed (Participants) | 20 | 20
percentage of oxygen saturation | 98.6 (2.1) | 98.5 (2.0)

4. Secondary Outcome: Pain Intensity on an 11-point Scale in the Postoperative Period
Description: The effect of low versus normal pCO2 concentrations on postoperative pain will be studied. Painscores are obtained at 15 minutes intervals and are expressed as a number on a 10 point scale (numeric rating scale; 1 (low)-10(maximum)). The data is avaraged over time
Time Frame: from the end of surgery untill 2 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypocapnia | Normocapnia
Number analyzed (Participants) | 20 | 20
units on a scale | 4.1 (3.3) | 4.0 (3.1)

5. Secondary Outcome: Sedation
Description: The effect of low versus normal pCO2 concentrations on postoperative sedation will be studied using the using the validated Leiden Observer's Assessment of Alertness/Sedation (0 (awake) - 6 (unarousable)) scale at 15 min intervals. The data are averaged over time.
Time Frame: from the end of surgery untill 2 hours postoperative
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hypocapnia | Normocapnia
Number analyzed (Participants) | 20 | 20
units on a scale | 2.4 (0.9) | 2.3 (0.8)

6. Secondary Outcome: Nausea
Description: The effect of low versus normal pCO2 concentrations on the incidence of postoperative nausea will be studied. The incidence is expressed as the percentage of people experiencing nausea per arm.
Time Frame: from the end of surgery untill 2 hours postoperative
Measure: Number; unit: percentage of patients
Arm/Group | Hypocapnia | Normocapnia
Number analyzed (Participants) | 20 | 20
percentage of patients | 3.6 | 5.9

7. Secondary Outcome: Vomiting
Description: The effect of low versus normal pCO2 concentrations on the incidence of postoperative vomiting will be studied. The incidence of vomiting is expressed as a precentage of the patients per arm.
Time Frame: from the end of surgery untill 2 hours postoperative
Measure: Number; unit: percentage of patients
Arm/Group | Hypocapnia | Normocapnia
Number analyzed (Participants) | 20 | 20
percentage of patients | 0 | 3.9

ADVERSE EVENTS:
Arm/Group | Hypocapnia | Normocapnia
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No